CLINICAL TRIAL: NCT02243891
Title: Left Atrial Ablation for Paroxysmal Atrial Fibrillation and Hypertension With Implantable Loop Recorder With or Without ROX Coupler Follow Up Study: The LAAPITUP 3 Study
Brief Title: AF Ablation With or Without ROX Coupler Study
Acronym: LAAPITUP3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neil Sulke (Other)
Responsible Party: Sponsor-Investigator, Neil Sulke, Consultant Cardiologist, Eastbourne General Hospital
Organization: Eastbourne General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAAPITUP3
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Atrial Fibrillation; Hypertension
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Atrial fibrillation ablation only
  Interventions: Procedure: Atrial fibrillation ablation
- ROX Coupler (Experimental): Atrial fibrillation ablation with concurrent ROX Coupler insertion
  Interventions: Procedure: Atrial fibrillation ablation; Procedure: ROX Coupler insertion

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Percutaneous catheter ablation for Atrial fibrillation.
Procedure: ROX Coupler insertion — The ROX Coupler is a CE-marked device designed to maintain an iliac arteriovenous fistula
  Arms: ROX Coupler

SUMMARY:
The study will test the hypothesis that ablation of paroxysmal atrial fibrillation in hypertensive subjects is more effective when a ROX coupler is inserted concurrently.

DETAILED DESCRIPTION:
The single blinded, randomised study is planned to commence in October 2014 after obtaining Research Ethics Committee and NHS Research and Development approval. A target of 20 participants with symptomatic paroxysmal AF will be recruited. All participants will be blinded and randomised to AF ablation only or AF ablation + ROX coupler implant. All participants will have right and left heart catheterisation prior to AF ablation +/- ROX coupler insertion. Participants will be followed up 6 weeks, 3, 6 months and 12 months after the ablation. The study will take place at Eastbourne District General. The study duration per patient is 13months. The overall study duration will be 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal AF suitable for AF ablation.
* Office Systolic blood pressure ≥ 140 mmHg based on an average of 3 blood pressure readings
* Ambulatory Blood Pressure Monitoring (ABPM) daytime average systolic blood pressure (SBP) ≥ 135 mmHg;
* Resistant Hypertension: Patients with established hypertension (diagnosed ≥ 12 months prior to baseline) and is on a guideline based drug regimen at a stable and a fully tolerated dose, consisting of ≥3 hypertensive medications (including 1 diuretic), or
* Uncontrolled Hypertension: Patient has drug intolerances to antihypertensive medications and is unable to take a guideline based drug regimen
* VO2 peak > 15mls/Kg/min on Cardiopulmonary exercise testing (CPX)
* Peak RER > 1.0 on Cardiopulmonary exercise testing
* Age over 18 years old.
* Informed consent to participate in this study.

Exclusion Criteria:

* Secondary hypertension amenable to conventional therapy
* Left ventricular systolic dysfunction with EF < 50%
* E/E' > 15 on transthoracic echocardiography
* Uncontrolled diabetes.
* Body Mass Index > 40 kg/m2
* Contraindicated for treatment with an arteriovenous anastomosis or interventional vascular procedure
* Severe chronic kidney disease as indicated by estimated glomerular filtration rate < 30 mL/min/1.73m2 using the MDRD calculation
* Renal denervation within the last 6 months
* Significant peripheral arterial and/or venous disease in the lower limbs (including unprovoked deep vein thrombosis, significant lower extremity edema and/or venous insufficiency)
* Current diagnosis of unstable cardiac disease requiring intervention,or significant history of serious cardiac comorbidity that may affect patient safety or study outcomes
* Current diagnosis of severe cerebrovascular disease or stroke within the past year
* Female patient who is pregnant, breastfeeding or planning to become pregnant; females of child-bearing potential must have a negative urine pregnancy test prior to treatment
* Any known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements
* Scheduled or planned surgery in the next 6 months that may affect patient safety or study outcomes
* Concurrent enrollment in another clinical trial without prior approval of ROX Medical, Inc.
* Any serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the study, comply with follow-up requirements or impact the scientific integrity of the study
* Intolerant or allergic to all anti-thrombolytic medications including aspirin
* Pulmonary arterial hypertension (PAH) defined as mean pulmonary artery pressure (mPAP) >30 mmHg as measured by right heart catheterization
* Pulmonary capillary wedge pressure (PCWP) > 15mmHg as measured by right heart catheterization
* Pre-existing ILRs or permanent pacemakers that do not allow for continuous monitoring for AF occurrence.
* Participation in a conflicting study.
* Potential participants who are mentally incapacitated and cannot consent or comply with follow-up.
* Pregnancy.
* Other cardiac rhythm disorders.
* Severe aortic and mitral valve disease.
* Previous ROX coupler implantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
AF ablation success | 3 months
  No AF burden detected on implantable loop recorder

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sulke, DM, Principal Investigator — East Sussex healthcare NHS trust
Locations (1):
- Eastbourne District General Hospital, Eastbourne, East Sussex, United Kingdom